CLINICAL TRIAL: NCT07287488
Title: Development and Evaluation of an Innovative Urethral Catheter Traction Device for Hemorrhage Control Following Transurethral Resection of the Prostate (TURP)
Brief Title: Development and Pilot Evaluation of a Urethral Catheter Traction Device for Post-TURP Hemorrhage Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Özlem Yılmaz, PhD Student / Doctoral Candidate (Clinical Nurse Specialist background), Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: AEŞH-EK-2025-218
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Simulation Study on Urethral Catheter Traction for Postoperative Hemorrhage Control After TURP
Keywords: TURP (Transurethral Resection of Prostate); Urethral Catheter Traction; Bleeding Control in TURP; Catheter Traction Techniques

STUDY DESIGN:
Intervention Model Description: Randomized Crossover Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The intervention was tested on mannequins; users and investigators were aware of the intervention, but outcome assessment was blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants apply the innovative urethral catheter traction device on mannequins. Post-procedure, users complete the "Catheter Traction Procedure Evaluation Form" and the Quebec Assistive Technology User Satisfaction Survey.
  Interventions: Device: Innovative Urethral Catheter Traction Device
- Control Arm (Active Comparator): Participants perform routine urethral catheter traction application on mannequins. Post-procedure, users complete the "Catheter Traction Procedure Evaluation Form".
  Interventions: Procedure: Routine Urethral Catheter Traction

INTERVENTIONS:
Device: Innovative Urethral Catheter Traction Device — A prototype urethral catheter traction device applied on mannequins to assess usability, safety, and effectiveness. Participants (operating room nurses and urology physicians) apply the device following a standardized protocol. Outcome assessment is performed by blinded assessors. Post-procedure, participants complete evaluation forms and user satisfaction surveys.
  Arms: Intervention Arm
Procedure: Routine Urethral Catheter Traction — Standard catheter traction method performed on mannequins, representing usual clinical practice. Participants apply traction according to routine procedures. Outcome assessment is performed by blinded assessors. Post-procedure, participants complete evaluation forms.
  Arms: Control Arm

SUMMARY:
Benign prostatic hyperplasia (BPH) is a common condition among elderly men. Transurethral resection of the prostate (TURP) is the gold standard surgical procedure, but postoperative bleeding is a frequent complication. Traditional catheter traction methods to control bleeding-such as fixing the catheter to the thigh or abdomen or using weights-have limitations, including restricted patient mobility, inconsistent pressure, and risk of infection or irritation.

This study aims to develop an innovative urethral catheter traction device that provides effective and stable pressure, is easy to apply, and minimizes potential complications. The device was tested in a simulated environment on mannequins. Both users and investigators were aware of the intervention, while outcome assessment was blinded. The study also evaluates healthcare professionals' perspectives on the usability, safety, and practicality of the device.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common health issue among elderly men, and transurethral resection of the prostate (TURP) is the gold standard surgical intervention. Postoperative bleeding is one of the most frequent complications of TURP, and controlling hemorrhage is essential for patient safety. Traditional methods for applying traction to the urethral catheter, including fixing the catheter to the thigh or abdomen or attaching weights to the catheter tip, have demonstrated efficacy in bleeding control. However, these approaches have several significant drawbacks:

* Restricted patient mobility, which may increase the risk of deep vein thrombosis (DVT)
* Inconsistent pressure on the prostatic capsule due to patient movement
* Risk of infection if materials become wet
* Irritation and discomfort due to friction on the glans penis
* Difficulty maintaining consistent and sustainable traction In clinical practice, an alternative method often used involves securing the catheter with gauze around the penis after applying traction. While this method allows patient mobility, it still carries risks related to hygiene, durability, and discomfort.

Given these limitations, there is a need for a device that can provide effective, stable, and safe traction, while being easy to apply and comfortable for the patient.

This study focuses on the development and evaluation of an innovative urethral catheter traction device. The device was tested in a simulated environment using mannequins. The intervention was fully visible to both the users and investigators, ensuring proper handling and application, while outcome assessment was conducted in a blinded manner to reduce bias.

The primary objectives of this study are:

1. To assess the usability and practicality of the new catheter traction device in a simulated environment
2. To evaluate healthcare professionals' perspectives regarding the safety, effectiveness, and ease of application of the device This study provides essential preliminary data for the design of future clinical trials involving human participants, aiming to improve postoperative hemorrhage management following TURP.

ELIGIBILITY:
Inclusion Criteria:

* Active operating room nurse or urology specialist physician.
* Experienced in urethral catheter application.
* Signed informed consent form voluntarily.

Exclusion Criteria:

* Individuals who do not wish to participate or withdraw consent during the study.
* Individuals who do not meet the inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Ease of Application Between the Innovative and Routine Urethral Catheter Traction Methods | Immediately after each intervention session (within 1 hour).
  This outcome assesses the ease of application of the newly developed urethral catheter traction device compared to the traditional traction method during simulated practice on mannequins. Participants will rate ease of use based on a standardized "Urethral Catheter Traction Procedure Evaluation Form." Related Hypothesis (H₁₀): There is no significant difference in ease of application between the innovative device and the traditional method.

SECONDARY OUTCOMES:
Stability and Safety of Catheter Traction Between the Innovative and Routine Methods | Immediately after both intervention and control sessions.
  This outcome evaluates the stability and safety of catheter traction provided by the innovative device compared with the routine method. Participants and assessors will evaluate tractive stability and potential complications (e.g., displacement, pressure inconsistency) using structured observation checklists.
  Related Hypothesis (H₂₀): There is no significant difference in stability and safety of traction between the innovative device and the traditional method.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik Şehir Hastanesi, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, individual participant data will not be shared. Data are limited and anonymized.